CLINICAL TRIAL: NCT05663944
Title: REpurposing SirolimUS in Compensated Advanced Chronic Liver Disease. the RESUS Proof of Concept Study
Acronym: RESUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20GA057
Record Dates: First submitted 2022-10-19; First posted 2022-12-23 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Advanced Chronic Liver Disease
Keywords: mTOR; liver fibrosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Randomised, patient-blinded, placebo-controlled, proof of concept, parallel group, single centre trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomised to sirolimus or placebo. To ensure reasonable costs at this early stage of study, the placebo will not be identically matched. The participants and their clinical care providers will be blinded. In this proof of concept study, sirolimus is not expected to have a recognisable health benefit to the participants and therefore unlikely to lead to unblinding of allocated treatment. Further, blinding will be maintained throughout the trial by having random titration schedules in the placebo arm. The Investigating team and pharmacy representative will not be blinded at this early stage of study. The final unblinding of all trial participants will be undertaken after the creation of a locked analysis data set.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 15 participants will receive a non-identical placebo tablet. They will be asked to take the placebo daily, exactly as instructed for the intervention arm, be subject to monitoring and random titration to mirror the study drug
  Interventions: Diagnostic Test: 1st MRI scan; Procedure: 1st Percutaneous or Endoscopic Ultrasound guided liver biopsy; Drug: Placebo 0.5mg capsule; Diagnostic Test: Baseline Blood Tests; Diagnostic Test: Baseline Clinical Examination; Diagnostic Test: Week 1 - 5 Titration Blood Tests; Other: Month 2 Clinical Examination; Diagnostic Test: Month 2 Blood Tests; Other: Month 4 Clinical Examination; Diagnostic Test: Month 4 Blood Tests; Other: Month 6 Clinical Examination; Diagnostic Test: Month 6 Blood Tests; Procedure: 2nd Percutaneous or Endoscopic Ultrasound guided liver biopsy
- Sirolimus (Experimental): 30 participants will be randomised to the study drug.
  Interventions: Drug: Sirolimus 0.5Mg Tab; Diagnostic Test: 1st MRI scan; Procedure: 1st Percutaneous or Endoscopic Ultrasound guided liver biopsy; Diagnostic Test: Baseline Blood Tests; Diagnostic Test: Baseline Clinical Examination; Diagnostic Test: Week 1 - 5 Titration Blood Tests; Other: Month 2 Clinical Examination; Diagnostic Test: Month 2 Blood Tests; Other: Month 4 Clinical Examination; Diagnostic Test: Month 4 Blood Tests; Other: Month 6 Clinical Examination; Diagnostic Test: Month 6 Blood Tests; Procedure: 2nd Percutaneous or Endoscopic Ultrasound guided liver biopsy

INTERVENTIONS:
Drug: Sirolimus 0.5Mg Tab — Once randomised, participants will receive either sirolimus or placebo daily for 6 months. Participants will start on a dose of 1mg daily (2 x 0.5mg tablets) and will have weekly routine bloods including full blood count, renal function and electrolytes and liver function test along with sirolimus trough levels measured to determine the next dose. The aim will be to achieve a steady state blood trough level of 3-7 ng/ml, which is usually achieved in 3-5 weeks. Placebo will also be started at 2 capsules daily. All participants will undergo weekly blood tests for the first 3-5 weeks and placebo doses will be adjusted randomly to maintain blinding.
  All participants will be reviewed by a research clinician at 2, 4 and 6 months.
  Other Names: Rapamycin
  Arms: Sirolimus
Diagnostic Test: 1st MRI scan — If participants opt in for MRI scans, a non-contrast MRI scan will be undertaken at Sir Peter Mansfield Imaging Centre, University of Nottingham at the start of the trial, and at the end, after 6 months of taking trial medication. This is to see whether any radiological features of fibrosis change can be detected to correlate with histological findings.
Procedure: 1st Percutaneous or Endoscopic Ultrasound guided liver biopsy — After informed consent, participants will undertake up to a 8-week screening period to provide baseline data to ensure eligibility. During this period, participants will undergo blood tests, percutaneous or endoscopic ultrasound-guided liver biopsy, unless the participant has undergone a liver biopsy within the past 3 months, in which case the previous liver biopsy sample will be utilised for this study. They will undergo a second liver biopsy at the end of the study, after taking 6 months of the study drug, to look for any histological change in fibrosis progression rate with sirolimus when compared to placebo
Drug: Placebo 0.5mg capsule — Once randomised, participants will receive either sirolimus or placebo daily for 6 months. The placebo is unmatched. Participants will start on a dose of 1mg daily (2 x 0.5mg capsules) and will have weekly routine bloods including full blood count, renal function and electrolytes and liver function test along with sirolimus trough levels, to maintain blinding of the research team members carrying out blood tests. Placebo doses will be adjusted randomly, in a pattern that mirrors the adjustments made to participants on sirolimus.
  All participants will be reviewed by a research clinician at 2, 4 and 6 months.
  Other Names: Placebo
  Arms: Placebo
Diagnostic Test: Baseline Blood Tests — During the initial clinical visit, venous blood samples will be taken to ensure that participants have no significant organ dysfunction:
  * Full blood count
  * Urea and electrolytes
  * Liver function tests
  * Clotting screen
  Research bloods will also be taken:
  - 5ml EDTA blood for storage and subsequent fibrosis marker analysis once all participants have complete study
Diagnostic Test: Baseline Clinical Examination — A thorough medical examination will be undertaken at the first clinical visit (cardiovascular, respiratory, abdominal, neurological, musculoskeletal, skin), to ensure participants are clinical stable. This will also serve as a comparator for future clinical examinations once participants have commenced the study drug.
Diagnostic Test: Week 1 - 5 Titration Blood Tests — Participants will start on a dose of 1mg daily (2 x 0.5mg tablets) and will have weekly bloods:
  * full blood count,
  * urea and electrolytes and
  * liver function tests to check the study drug is not causing any significant organ damage.
  * Sirolimus trough levels will be measured to determine the next dose. The aim will be to achieve a steady state blood trough level of 3-7 ng/ml, which is usually achieved in 3-5 weeks. Therefore, participants will have a minimum of 3 weeks of blood tests during this period, The need for week 4 and 5 blood tests will be decided by the trial pharmacist who will be monitoring results.
  Placebo will also be started at 2 capsules daily. All participants will undergo weekly blood tests for the first 3-5 weeks and placebo doses will be adjusted randomly to maintain blinding.
Other: Month 2 Clinical Examination — A thorough medical examination will be undertaken at Month 2 (cardiovascular, respiratory, abdominal, neurological, musculoskeletal, skin), to ensure participants remain clinically stable whilst on the study drug. They will also be asked about potential side effects in detail.
Diagnostic Test: Month 2 Blood Tests — During the Month 2 clinical visit, venous blood samples will be taken to ensure that participants have no significant organ dysfunction:
  * Full blood count
  * Urea and electrolytes
  * Liver function tests
  * Clotting screen
  * Sirolimus trough level will also be repeated to ensure that the previously titrated study drug has remained in steady state
  Research bloods will also be taken:
  - 5ml EDTA blood for storage and subsequent fibrosis marker analysis once all participants have complete study
Other: Month 4 Clinical Examination — A thorough medical examination will be undertaken at Month 4 (cardiovascular, respiratory, abdominal, neurological, musculoskeletal, skin), to ensure participants remain clinically stable whilst on the study drug. They will also be asked about potential side effects in detail.
Diagnostic Test: Month 4 Blood Tests — During the Month 4 clinical visit, venous blood samples will be taken to ensure that participants have no significant organ dysfunction:
  * Full blood count
  * Urea and electrolytes
  * Liver function tests
  * Clotting screen
  * Sirolimus trough level will also be repeated to ensure that the previously titrated study drug has remained in steady state
  Research bloods will also be taken:
  - 5ml EDTA blood for storage and subsequent fibrosis marker analysis once all participants have complete study
Other: Month 6 Clinical Examination — A thorough medical examination will be undertaken at Month 6 (cardiovascular, respiratory, abdominal, neurological, musculoskeletal, skin), to ensure participants have remained clinically stable whilst on the study drug. At this visit, they will be asked to finish taking the study drug. They will also be asked about potential side effects in detail.
Diagnostic Test: Month 6 Blood Tests — During the Month 6 clinical visit, venous blood samples will be taken to ensure that participants have no significant organ dysfunction:
  * Full blood count
  * Urea and electrolytes
  * Liver function tests
  * Clotting screen
  * Sirolimus trough level will also be repeated to ensure that the previously titrated study drug has remained in steady state
  Research bloods will also be taken:
  - 5ml EDTA blood for storage and subsequent fibrosis marker analysis once all participants have complete study
Procedure: 2nd Percutaneous or Endoscopic Ultrasound guided liver biopsy — All participants will undergo a second liver biopsy at the end of the study, after taking 6 months of the study drug, to look for any histological change in fibrosis progression rate when compared to their first biopsy.
Diagnostic Test: 1st MRI scan — If participants opt in for MRI scans, a non-contrast MRI scan will be repeated at the end of the trial, after 6 months of taking trial medication. This is to see whether any radiological features of fibrosis change can be detected to correlate with histological findings.

SUMMARY:
Background: Advanced liver scarring leads to liver failure, liver cancer and premature death. It mainly affects people in the working age group (18-65 years) and is the only major cause of death that is still increasing every year in the UK. It costs the NHS £2.1 billion a year. This will continue to rise due to increasing alcohol misuse and the obesity crisis.

Advanced liver scarring remains incurable as there is no treatment to slow progression of scarring. Sirolimus is a medication that has been used to prevent rejection after organ transplantation for over 20 years. It reduces liver scarring, improves liver functioning and prolongs life in animals. It has also been shown to reduce liver scarring in patients after liver transplantation. Sirolimus, therefore offers a potential treatment option for liver scarring.

Question and Objectives: If used in patients with advanced liver scarring, can sirolimus slow the progression of scarring? The main objective is to undertake a small-scale study (proof of concept) to investigate if sirolimus could slow the progression of scarring in patients with advanced liver scarring using clinically relevant biomarkers, which will see if the liver responds to treatment. How it will be done: The study will be conducted in Nottingham University Hospitals NHS Trust. 45 patients with advanced liver scarring will be randomly given either sirolimus or placebo tablets daily for 6 months. Participants will have a liver biopsy and a MRI scan at the start and end of the study to measure the change in the biomarkers of liver scarring. A reduction in these markers will indicate successful treatment. Participants will be monitored for safety of the drug. Potential Impact: If found efficacious, sirolimus would provide an acceptable treatment for patients with advanced liver scarring and would also save a substantial sum of money for the NHS.

DETAILED DESCRIPTION:
TRIAL DESIGN This is a phase II, randomised, patient-blinded, placebo-controlled, proof of concept, parallel group single centre trial. Phase I information is not required since sirolimus has been in use for other therapeutic indications.

STUDY SETTING This is a single centre study and will be undertaken at Nottingham University Hospitals NHS Trust.

TRIAL PROCEDURES Recruitment Recruitment will be over 15 months from hepatology clinics. Based on previous experience, recruiting 3 patients per month will achieve the recruitment of 45 participants over 15 months. Progression criteria around recruitment, retention and treatment compliance will be defined as assessed at three monthly intervals.

Patient identification The chief investigator who is part of the clinical team will identify potential participants by reviewing patient records (e.g., previous clinic letters) of patients attending hepatology clinics. Information packs (patient information sheet and trial team contact details) will be sent to all patients who appear to meet the eligibility criteria. A delegated research professional (e.g., research nurse) will then gauge the interest of the patient through a telephone call 1 - 2 weeks after sending the information pack via post.

Screening Screening will include a baseline clinic which will involve eligibility check, medical history and general physical examination, informed consent, routine bloods and liver biopsy, followed by an MRI scan 2 weeks after the baseline clinic visit.

Medical history will include clinically significant diseases, surgeries, reproductive status, smoking history, use of alcohol and illicit/recreational drugs and all medication (prescription and over the counter drugs, herbal and homeopathic remedies, nutritional supplements) used by the patient within 90 days prior to the baseline clinic visit. A full physical examination will include general, cardiorespiratory, abdominal and neurological examination. Routine bloods and a liver biopsy (either percutaneous or endoscopic ultrasound guided) will be performed, unless the participant has had a liver biopsy within the past 3 months of the baseline clinic visit. Participants will then undergo an optional MRI scan at Sir Peter Mansfield Imaging Centre, University of Nottingham 2 weeks after the baseline clinic. If participants are found to be ineligible using all criteria, clinical care will continue as usual. Anonymised information on participants who are not randomised will be kept for CONSORT reporting the generalisability of the results.

Consent Written informed consent for participation in the study will be obtained before performing any study-specific screening tests or evaluations. Written informed consent maybe obtained up to 28 Days before the start of the study. Informed consent forms for enrolled patients and for patients who are not subsequently enrolled will be maintained at the study site. A copy of signed consent form will be provided to the patient or their authorised representative. All signed and dated consent forms will remain in each patient's study file and will be available for verification at any time. The consent form will be revised if there are any changes to the study procedures or if new information becomes available that may affect the willingness of the patient to participate.

The randomisation scheme All screening evaluations will be completed and reviewed to confirm that patients meet all eligibility criteria before randomisation. A screening log will be maintained to record details of all patients screened and to confirm eligibility or record the reasons for the screening failure, as appropriate. Randomisation will be 2:1 (sirolimus:placebo) to allow interpretation of safety and provide an indication of placebo response for future trial development.

Baseline data After informed consent, participants will undertake up to a 4-week screening period to provide baseline data to ensure eligibility. During this period, participants will undergo blood tests, transjugular liver biopsy and MRI scan. At baseline clinic (visit 1), routine bloods including full blood count, electrolytes and renal function, liver function test, and clotting screen will be collected. Blood will also be collected for extraction of serum and plasma. A liver biopsy will be undertaken on the same day as the baseline clinic (visit 1), unless the participant has undergone a liver biopsy within the past 3 months, in which case the previous liver biopsy sample will be utilised for this study with the consent of the patient. A non-contrast MRI scan will be undertaken at Sir Peter Mansfield Imaging Centre, University of Nottingham 2 weeks after the baseline clinic/liver biopsy. Trial assessments Once randomised, participants will receive either sirolimus or placebo daily for 6 months. Participants will start on a dose of 1mg daily (2 x 0.5mg tablets) and will have weekly blood sirolimus trough levels measured to determine the next dose. The aim will be to achieve a steady state blood trough level of 3-7 ng/ml, which is usually achieved in 3-5 weeks. Placebo will also be started at 2 tablets daily. All participants will undergo weekly blood tests for the first 3-5 weeks and placebo doses will be adjusted randomly to maintain blinding. All participants will be reviewed by a research nurse at 2, 4 and 6 months (visits 3, 4 and 5) and the following will be recorded: assessment of toxicity of previous dose, weight, routine bloods - full blood count, electrolytes and renal function, liver function test and clotting screen, blood sirolimus trough levels and serum and plasma samples for research. Sirolimus dose will be adjusted according to the blood sirolimus trough level to maintain a blood trough level of 3- 7ng/ml, as needed. Measurement of sirolimus trough levels will also be used, along with tablet counting, to assess compliance. Only the trial pharmacist will be unblinded and involved in dose adjustment and tablet counting. They will liaise with the chief investigator if needed.

All participants will undergo a repeat liver biopsy at 6 months and a non-contrast MRI scan at the Sir Peter Mansfield Imaging Centre, University of Nottingham 2 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* capable of giving informed consent
* aged 18-75 years
* compensated advanced chronic liver disease (Child Pugh class A) due to excess alcohol consumption or fatty liver disease
* willing to and able to undergo percutaneous or endoscopic ultrasound-guided liver biopsy at baseline and at 6 months

Exclusion Criteria:

* inability to provide informed consent
* inability to comply with the study protocol
* subjects who may be unavailable for the duration of the treatment course, likely to be noncompliant, or who are felt to be unsuitable by the Investigator for any other reason
* previous history of decompensation of liver disease or liver cancer
* women who are pregnant or breastfeeding
* unable or unwilling to use highly effective contraception during and 12 weeks after the trial participation
* history of allergy or adverse event to sirolimus
* previous or current use of sirolimus
* concurrent use of experimental agents
* an unstable or uncontrolled medical disorder which in the investigator's opinion precludes recruitment within the trial
* major medical comorbidities (e.g., end-stage organ disease, cancer or immunodeficiency)
* increased risk of infectious complications (e.g., immunodeficiency, recent live vaccination)
* surgery within the past 6 months or an anticipated requirement for surgery during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
proportion of deactivation of activated HSCs from baseline to 6 months | 6 months
  The primary objective is to determine proportion of deactivation of activated HSCs by sirolimus compared to placebo, in patients with advanced chronic liver disease from baseline to 6 months. This will be measured by the change in the proportion in alpha smooth muscle actin (αSMA) expression in the liver biopsies at baseline and at 6 months in the sirolimus and placebo groups. Alpha smooth muscle actin is a protein present in fibrotic tissue. It is stained for during histological analysis. The presence of alpha smooth muscle actin is reported as a proportion of the tissue sample e.g., 60% of this tissue sample stained positively for alpha smooth muscle actin. Response to treatment is defined as a reduction in αSMA of at least 50% from baseline to 6 months e.g., now only 30% stains positive. It is impossible to say what the average starting proportion would be as this varies significantly from patient to patient. What is important is the proportionate change.

SECONDARY OUTCOMES:
change in histological fibrosis stage from baseline to 6 months | 6 months
  Change in histological fibrosis stage will be determined through change in collagen bundle morphology (descriptive terms: Collagen orientation ranges from perfectly random to perfectly parallel. Collagen bundle packing signifies the average distance between the centres of collagen bundles. Universally accepted visual patterns e.g. peri-cellular collagen bundles, bridging collagen bundles etc indicate fibrosis severity).
change in multiparametric MRI measures from baseline to 6 months | 6 months
  Changes in liver architecture will be measured using liver T1/T2/T2*, diffusion, and volume, and renal T1. T1 and T2 refer to the relaxation times used when scanning tissue as an interval between pulse sequences. The T1 technique regulates the rate that protons revert to their regular rotation, and T2 decides the rate at which protons achieve equilibrium or operate at different times. Creating T1 weighted images requires a short time to echo (TE) and repetition times (TR). These refer to the duration between the radiofrequency pulse's delivery and the capture of the echo signal, and the measured time between pulse sequences applied to an area, respectively. On the other hand, T2 weighted images use longer TE and TR times. A longer TE time would indicate a stiffer liver.
the safety and tolerability of sirolimus in patients with advanced chronic liver disease | 6 months
  Safety and tolerability will be monitored during clinic visits and through adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided